CLINICAL TRIAL: NCT00486395
Title: Offering Less Invasive Ventilation in Infants Born 28 to 32 Weeks Gestation: A Randomized Controlled Trial.
Brief Title: Will CPAP Reduce Length Of Respiratory Support In Premature Infants?
Acronym: OLIVIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decreasing recruitment
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Collaborators: Child and Family Research Institute (Other)
Responsible Party: Principal Investigator, Rebecca Sherlock, Neonatologist, Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-08 005
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Prematurity; Respiratory Distress Syndrome, Newborn
Keywords: prematurity; randomized trial; RDS; surfactant; CPAP; ventilation
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome, Newborn; Respiratory Aspiration | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Mechanical ventilation
  Interventions: Device: Mechanical ventilation
- 2 (Experimental): CPAP
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP administered via "Bubble" method or Infant Flow Driver
  Arms: 2
Device: Mechanical ventilation — Volume guarantee strategy
  Arms: 1

SUMMARY:
In Canada each year, there are approximately 800 infants born between 28 and 32 weeks gestation. Up to 60% of these infants will require breathing tube placement for Respiratory Distress Syndrome or RDS. RDS is a lung disease of prematurity due to a lack of a compound called surfactant. The breathing tube is placed as a conduit for placing surfactant into the babies' lungs to improve the lung disease. Most babies are then placed on a breathing machine or ventilator. Ventilation is not without harm and can be associated with lung damage, delays in feeding, increased hospital stay and interruption of bonding. An alternative that does not require the presence of a breathing tube is Continuous Positive Airway Pressure (CPAP). We will randomize babies to either ventilation or CPAP to try to minimize the length of time the baby is kept on respiratory support.

DETAILED DESCRIPTION:
Objectives: To determine whether infants 28 to 32 weeks gestational age with RDS treated with surfactant followed by CPAP have a shorter length of respiratory support (length of time on a ventilator and CPAP) than similar infants who are treated with MV after surfactant therapy; and to examine secondary outcomes including outcomes related to lung disease, feeding issues and hospital length of stay (secondary outcomes).

Hypothesis: The use of CPAP after surfactant in infants born 28 to 32 weeks with RDS will reduce the length of respiratory support as compared with infants treated with MV. We hypothesize that the incidence of lung disease and feeding issues will be similar between groups while length of hospital stay will be shorter in the CPAP group.

Methods: A multi-center, randomized trial conducted in seven neonatal intensive care units in Canada and France. Parents will be approached for consent prior to delivery or after the infant shows signs of RDS. Infants 28 to 32 weeks gestation with RDS will be eligible for the study. After intubation and surfactant administration, babies will be randomized to either receive CPAP or MV. Strict criteria for CPAP failure, weaning ventilation and weaning and discontinuing CPAP will be specified. Infants will be followed in the nursery until hospital discharge or until all outcomes have been determined.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born greater than or equal to 28 weeks (28+0) and less than 32 weeks (31+6) gestation admitted to the NICU at a participating center
2. Diagnosis of RDS in the first 24 hours of life requiring intubation for surfactant administration by any combination of the following: Classic clinical signs of RDS include tachypnea, moderate to severe intercostal and subcostal retractions, grunting respirations and oxygen needs of >0.30 and/or on CPAP of 5 to 6 H2O cm and/or radiographic signs of RDS including low lung volumes, a reticular-granular pattern of lung infiltrates and air bronchograms. A chest radiograph is not a mandatory criterion for the diagnosis of RDS if clinical signs are present
3. Parental consent obtained.

Exclusion Criteria:

1. Infants with a major congenital anomaly
2. Infants with pulmonary hypoplasia; 3. Infants known or suspected to have a neuromuscular disorder;
3. Infants from mothers that had greater than 2 weeks ruptured membranes.
4. Infants that had vigourous resuscitation including chest compressions and cardiac meds.
5. No parental consent obtained.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Length of respiratory support | Variable
  CPAP plus MV days

SECONDARY OUTCOMES:
Duration of ventilation, duration of oxygen therapy, pneumothorax rate and BPD by Walsh test, time to full feeds, time to regain birthweight, necrotizing enterocolitis, time to discharge, achievement of readiness for discharge criteria | Variable

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Sherlock, MD, FRCPC, PhD(c), Principal Investigator — Children's and Women's Health Centre of BC
Locations (6):
- Canada (6):
  - The Royal Alexandra Hspital, Edmonton, Alberta
  - The Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Children's and Women's Health Centre of BC, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - The Ottawa Hospital-General campus, Ottawa, Ontario